CLINICAL TRIAL: NCT06318858
Title: Efficacy of Daily and Weekly Iron Supplementation on Anemia Prevalence in Thai Infants Aged 6-12 Months
Brief Title: Daily and Weekly Iron Supplementation in Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Suranaree University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MU-CIRB 2022/313.1411
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Anemia; Iron Status; Infants; Iron
Keywords: Anemia; Iron status; Infants; Iron supplementation
MeSH Terms: conditions — Anemia | interventions — Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: group 1: daily iron syrup supplementation group 2: weekly iron syrup supplementation
Who Masked: Participant, Care Provider, Investigator
Masking Description: Letter codes were assigned to the iron syrup and the placebo by researchers who have not involved in the study. The codes have been kept until data analysis and report writing are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 daily iron supplementation (Experimental): 12.5 mg daily iron syrup supplementation from 6-9 months old, followed by 12.5 mg weekly iron syrup supplementation from 9-12 months old.
  Infants aged 6-9 months will receive two iron syrup bottles. One bottle aims for ingestion every Monday of the week, and one bottle aims for ingestion on other days of the week.
  At ages 9-12 months, infants will receive an iron syrup bottle that aims for ingestion every Monday of the week.
  Interventions: Dietary Supplement: Iron supplement
- Group 2 weekly iron supplementation (Other): 12.5 mg weekly iron syrup supplementation from 6-12 months old. Infants aged 6-9 months will receive an iron syrup bottle that aims for ingestion every Monday of the week and a placebo bottle that aims for ingestion on other days of the week.
  At ages 9-12 months, infants will receive an iron syrup bottle that aims for ingestion every Monday of the week.
  Interventions: Dietary Supplement: Iron supplement

INTERVENTIONS:
Dietary Supplement: Iron supplement — Group 1: 12.5 mg daily iron syrup supplementation from 6-9 months old

SUMMARY:
This study aims to compare the efficacy of daily iron supplementation and weekly iron supplementation in infants aged 6-12 months on the prevalence of anemia, hemoglobin level, and serum ferritin levels. Infants will be enrolled at 6 months and will be randomly assigned to receive either daily or weekly iron supplementation for the first 3 months and will be followed by weekly iron supplementation for another 3 months.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of daily iron supplementation and weekly iron supplementation in infants aged 6-12 months on the prevalence of anemia, hemoglobin level, and serum ferritin levels. Normal birth weight and term infants will be enrolled at 6 months based on the inclusion criteria. Eligible participants will be assessed at baseline, including anthropometry, dietary intake, and biochemistry (hemoglobin, iron status, vitamin A status, and inflammation). Participants will then be randomly assigned to receive either daily or weekly iron supplementation for the first 3 months. Participants will be followed up at 9 months for the same assessments and will receive weekly iron supplementation for another 3 months. Participants will be followed up at 12 months and the same assessments will be performed. After that, participants will go back to the routine health care service, weekly iron supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy infant, aged 6 months ± 2 weeks
* Having a birth weight between 2,500 and 4,000 grams
* Being born full term (37 to 41 weeks of age + 6 days)
* Having hemoglobin ≥ 10.5 g/dL
* Being planned to breastfeed with complementary food and/or complementary foods with formula milk

Exclusion Criteria:

* Infants with chronic illnesses or thalassemia clinical signs such as anemia, enlarged liver, or spleen (if parental history suggests the child is at risk of developing a thalassemia disease that may not show clinical symptoms)
* Previously or currently taking an iron supplement

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-08-14 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
Anemia status | at aged 6, 9, and 12 months
  Hemoglobin concentration will be assessed and classified as anemia or non-anemia.
Iron status | at aged 6, 9, and 12 months
  Serum ferritin will be assessed to reflect iron status

SECONDARY OUTCOMES:
Weight | at aged 6, 9, and 12 months
  Body weight will be assessed, and weight-for-age and weight-for-length Z scores will be generated
Length | at aged 6, 9, and 12 months
  Length will be assessed, and length-for-age Z scores and weight-for-length will be generated
Dietary intake | at aged 6, 9, and 12 months
  Dietary intake will be assessed using the 24-hr dietary recall for 3 days
Head circumference (HC) | at aged 6, 9, and 12 months
  HC will be assessed, and head circumference-for-age Z scores will be generated

OTHER OUTCOMES:
Hemoglobin typing | at aged 12 months
  Hemoglobin typing will be assessed
C-reactive protein (CRP) | at aged 6, 9, and 12 months
  High sensitivity CRP will be analyzed and will be used for the adjustment of serum ferritin
Alpha-1 acid glycoprotein (AGP) | at aged 6, 9, and 12 months
  AGP will be analyzed and will be used for the adjustment of serum ferritin
Serum transferrin receptor | at aged 6, 9, and 12 months
  Serum transferrin receptor will be assessed to reflect iron status
Serum Retinol Binding Protein (RBP) | at aged 6, 9, and 12 months
  RBP will be assessed to reflect vitamin A status

CONTACTS AND LOCATIONS:
Overall Officials: Tippawan Pongcharoen, PhD, Principal Investigator — Mahidol University
Locations (1):
- Samphran District Hospital, Sam Phran, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No